CLINICAL TRIAL: NCT00499213
Title: Home Care Assisted Peritoneal Dialysis: The Impact of Expanding Eligibility for Peritoneal Dialysis on Rates of Hospitalization
Brief Title: Rates of Hospitalization in Home Care Assisted Peritoneal Dialysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: London Health Sciences Centre (Other)
Other Study IDs: 07-22
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-07

CONDITIONS: Rate of Hospitalization

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Home Care Assisted Peritoneal Dialysis

SUMMARY:
We have developed and implemented a program that offers home care assistance to patients wishing to perform home peritoneal dialysis, but are unable to do it for themselves. This study is being conducted to ensure the safety of this dialysis program and specifically, to see if the risk of being hospitalized is increased when this therapy is provided to patients.

DETAILED DESCRIPTION:
The cost of caring for patients with kidney failure is growing at an alarming rate and accounts for up to 7% of health care expenditures in developed countries. The majority of the cost is due to in-centre hemodialysis (HD) because of high operating costs and the capital investment required to build new dialysis units. In recent years, there has been a shortage of in-centre HD beds and it has become a priority to increase the number of patients being treated in their place of residence with therapies like peritoneal dialysis (PD). Unfortunately, many patients are unable to perform their own dialysis at home, a trend that will become more and more common as the population ages. We developed and implemented a program of home care assisted PD at Sunnybrook Health Sciences Centre where health care workers go into the home to assist patients with their treatment. The program has been a success and has garnered national attention. As a result, it has been adopted province-wide as part of the "Provincial PD Joint Initiative" and the Manitoba Renal Program is currently implementing a similar program to increase the use of PD.

However, based on preliminary data, we are concerned that patients treated with home care assisted PD may have higher rates of hospitalization when compared to traditional forms of treatment (23.5 days per year of follow-up compared to 13 days per year of follow-up. If this is true it could have a significant impact on patient quality-of-life, cost-savings associated with PD, and resource allocation and planning in regional dialysis programs. This is of particular concern given that the provincial initiative has a goal of increasing the proportion of patients being treated with PD from the current 18% to 30% by 2010.

The primary objective of this study is to determine if patients treated with home care assisted peritoneal dialysis are more likely to be hospitalized when compared to those treated with in-centre hemodialysis.

The secondary objective of this study is to compare the occurrence of important outcome events including the need for access-related procedures, technique survival, and death in patients on home care assisted peritoneal dialysis compared to in-centre hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. End-stage kidney disease in the opinion of the attending nephrologist
3. Deemed eligible for both home assisted PD and traditional in-centre HD following a multidisciplinary assessment, regardless of what therapy is chosen

Exclusion Criteria:

1. History of kidney transplant or expected to receive a transplant in the next 3 months
2. Expected to transfer to another regional dialysis program following the initiation of dialysis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Quinn, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Matthew J Oliver, MD, MHS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada